CLINICAL TRIAL: NCT04566393
Title: Expanded Access to Ulixertinib (BVD-523) in Patients With Advanced MAPK Pathway-Altered Malignancies
Status: Available | Type: Expanded Access
Sponsor: xCures (Industry)
Collaborators: Cancer Commons (Other)
Responsible Party: Sponsor
Other Study IDs: ULI-EAP-100
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Cancer; Small Bowel Cancer; Colorectal Cancer; Melanoma; Non Small Cell Lung Cancer; Thyroid Cancer; Bladder Cancer; Head and Neck Cancer; Gastric Cancer; Esophageal Cancer; Cholangiocarcinoma; Ovarian Cancer; Hepatocellular Carcinoma; Glioblastoma; MAPK Gene Mutation; KRAS Activating Mutation; BRAF Gene Mutation; NRAS Gene Mutation; HRAS Gene Mutation; MEK Mutation; ERK Mutation
MeSH Terms: conditions — Pancreatic Neoplasms; Colorectal Neoplasms; Melanoma; Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms; Urinary Bladder Neoplasms; Head and Neck Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Cholangiocarcinoma; Ovarian Neoplasms; Carcinoma, Hepatocellular; Glioblastoma | interventions — ulixertinib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Ulixertinib (BVD-523) — Ulixertinib (BVD-523) is an oral, first-in-class ERK1/2 inhibitor

SUMMARY:
The objective of this expanded access program is to provide ulixertinib (BVD-523) for compassionate use in advanced cancer patients with MAPK pathway-altered solid tumor(s), including but not limited to KRAS, NRAS, HRAS, BRAF, MEK, and ERK mutations who have incomplete response to or have exhausted available therapies.

Ulixertinib is available for treatment as monotherapy or in combination with other clinically tolerable agent(s), conditionally approved by the drug manufacturer.

ELIGIBILITY:
Inclusion Criteria:

* Main Inclusion Criterion:

  1. Patient has a MAPK pathway-altered solid tumor(s), including but not limited to KRAS, NRAS, HRAS, BRAF, MEK, and ERK mutations.
* Other Inclusion Criteria:

  1. In the opinion of the treating physician, the patient has exhausted or has inadequate response to available anti-cancer treatments.
  2. In the opinion of the treating physician, the patient has adequate organ function to tolerate ulixertinib as defined in section 6.1
  3. Male or female patients aged ≥ 12 years.
  4. Patient must be able to swallow and retain orally administered medication.

     Note: Ulixertinib is primarily absorbed in the duodenum and therefore patients with any prior stomach or duodenal resection should be evaluated with that understanding.
  5. For females, evidence of post-menopausal status or negative urinary or serum pregnancy test for pre-menopausal patients.
  6. Highly effective contraception for both male and female patients throughout the treatment and for at least 4 months after last treatment administration. In patients under the age of 18, who are not sexually active, abstinence is an acceptable form.
  7. Toxicities related to any prior treatments are either stable, stable on supportive therapy, resolved, or in the opinion of the treating physician, clinically non-significant
  8. Ability to understand a written informed consent document, and the willingness to sign it. Assent will be obtained when appropriate based on the patient's age.

Exclusion Criteria:

1. Patient is already participating in or qualifies for and is able to enroll in a clinical trial of ulixertinib (BVD-523).
2. Patient has received systemic therapy with an investigational agent within 5 half-lives or 14 days prior to starting ulixertinib treatment, whichever is shorter.
3. Patient has received radiotherapy within 14 days prior to the first dose of ulixertinib treatment other than for the allowable treatment of symptomatic bone metastasis.
4. A history of current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR)
5. Current evidence of uncontrolled, significant intercurrent illness that would, in the treating physician's judgment, contraindicate the patient's treatment with ulixertinib due to safety concerns.
6. Patients who, in the opinion of the treating physician, have not fully recovered from recent major surgery to a sufficient extent to tolerate treatment with ulixertinib.
7. Known hypersensitivity to ulixertinib or any component in its formulation.
8. Patients taking prohibited medications as described in current Investigator's Brochure.

   Note: Patients who require treatment with Drugs that are strong inhibitors or inducers of CYP1A2, CYP2D6, and CYP3A4 (see Appendix 3) were excluded from the FIH study of ulixertinib and should be discussed with xCures to review if any potential benefits outweigh the potential risks.
9. Patient is actively breastfeeding.
10. Prior stomach or duodenal resection that in the opinion of the treating physician would affect the breakdown and absorption of ulixertinib.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Infirmary Cancer Care, Mobile, Alabama
  - PCR Oncology, Arroyo Grande, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - xCures Inc., San Francisco, California
  - Providence Saint John's Health Center, Santa Monica, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Orlando Health, Orlando, Florida
  - Mercy Medical Center, Cedar Rapids, Iowa
  - Unity Point Health - St. Lukes Hospital, Cedar Rapids, Iowa
  - Our Lady of the Lake Hospital, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Oakland Macomb Cancer Specialists, Sterling Heights, Michigan
  - Lake Region Healthcare, Fergus Falls, Minnesota
  - Nebraska Hematology Oncology, Lincoln, Nebraska
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Hunterdon Hematology Oncology, Flemington, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - The Minniti Center for Medical Oncology and Hematology, Mickleton, New Jersey
  - Atlantic Health System/Overlook Medical Center, Summit, New Jersey
  - Hirschfeld Oncology, Brooklyn, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - The Christ Hospital, Cincinnati, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania
  - MD Anderson, Houston, Texas
  - UTHealth Houston, Houston, Texas
  - UTHealth - Tyler, Tyler, Texas